CLINICAL TRIAL: NCT05393908
Title: Intraoperative Surgeon Administered Transversus Abdominis Plan (TAP) Block With Liposomal Bupivacaine and Post-operative Pain Control After Repeat Cesarean Delivery
Brief Title: Intraoperative TAP Block After Repeat Cesarean
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding became available for this study to be feasible
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Gianna Wilkie, Principal Investigator, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000407
Record Dates: First submitted 2022-05-18; First posted 2022-05-26 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Post-operative Pain
Keywords: Cesarean delivery, post-operative pain, TAP block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP Block Group (Active Comparator): Participants will receive a surgeon administered TAP block consisting of liposomal bupivacaine during their repeat cesarean delivery.
  Interventions: Procedure: TAP Block Group
- Standard of Care Postoperative Pain Control (No Intervention): Participants will not receive a surgeon administered TAP block consisting of liposomal bupivacaine during their repeat cesarean delivery and will receive the routine standard of care for post-operative pain control.

INTERVENTIONS:
Procedure: TAP Block Group — Participants will receive a surgeon administered TAP block.
  Arms: TAP Block Group

SUMMARY:
The aim of this study is to perform a randomized trial to investigate if intraoperative surgeon administered TAP block reduces pain and use of oral and parenteral pain medications after repeat cesarean delivery. The investigators aim to compare surgeon administered TAP block with liposomal bupivacaine compared to standard treatment (i.e. no TAP block) with regard to the primary outcome of post-operative narcotic use.

DETAILED DESCRIPTION:
Transversus abdominis plane (TAP) block is a well-described technique to provide a field block for analgesia. It has been shown to be effective in postoperative analgesia after cesarean delivery. TAP blocks are commonly performed post-operatively by anesthesiologists using liposomal bupivacaine with ultrasound guidance. Liposomal bupivacaine is an FDA approved medication for post-surgical analgesia and available at UMass-Memorial Medical Center. Liposomal bupivacaine provides sustained release of medication for up to 120 hours. A recent multicenter randomized controlled trial demonstrated the efficacy of anesthesiologist administered TAP blocks using liposomal bupivacaine after cesarean delivery. Infiltration of the skin and fascia with liposomal bupivacaine after cesarean did not have an effect and this can be explained by the path that the pain fibers take through the TAP which makes them amenable to a TAP block while a superficial infiltration is ineffective.The aim of this study is to perform a randomized trial to investigate if intraoperative surgeon administered TAP block reduces pain and use of oral and parenteral pain medications after repeat cesarean delivery. The investigators aim to compare surgeon administered TAP block with liposomal bupivacaine compared to standard treatment (i.e. no TAP block) with regard to the primary outcome of post-operative narcotic use.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women presenting for elective repeat cesarean delivery at 37-42 weeks gestational age.
* Pregnancy and delivery care obtained at UMass Memorial Medical Center
* Patients able to provide written informed consent
* English, Spanish, or Portuguese-speaking patients

Exclusion Criteria:

* Participants who are under the age of 18 years
* Active labor.
* Baseline pain score > 6.
* Unable to provide informed consent.
* Prisoners will be excluded from this research.
* Narcotic use in the 2 weeks prior to delivery.
* Active substance abuse.
* Inability to take narcotic analgesia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Daily Narcotic Use in Morphine Equivalents | From time of surgery through postpartum day 4
  Daily Narcotic Use in Morphine Equivalents

SECONDARY OUTCOMES:
Time to first administered narcotic (oral or parental) | From time of surgery through postpartum day 4
  Time to first administered narcotic (oral or parental) post cesarean delivery
Daily Average Pain Score | From time of surgery through postpartum day 4
  Daily Average Pain Score based on ten point pain scale (minimum 0, maximum 10) with higher numbers indicating worse pain
Daily Maximum Pain Score | From time of surgery through postpartum day 4
  Daily Average Pain Score based on ten point pain scale (minimum 0, maximum 10) with higher numbers indicating worse pain
Time to First Ambulation | From time of surgery through postpartum day 4
  Time to First Ambulation post cesarean delivery
Time to First Solid Food | From time of surgery through postpartum day 4
  Time to First Solid Food

CONTACTS AND LOCATIONS:
Overall Officials: Gianna Wilkie, MD, Principal Investigator — University of Massachusetts Chan Medical School

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilson RD, Caughey AB, Wood SL, Macones GA, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G. Guidelines for Antenatal and Preoperative care in Cesarean Delivery: Enhanced Recovery After Surgery Society Recommendations (Part 1). Am J Obstet Gynecol. 2018 Dec;219(6):523.e1-523.e15. doi: 10.1016/j.ajog.2018.09.015. Epub 2018 Sep 18. PMID 30240657
- [Background] Tsai HC, Yoshida T, Chuang TY, Yang SF, Chang CC, Yao HY, Tai YT, Lin JA, Chen KY. Transversus Abdominis Plane Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:8284363. doi: 10.1155/2017/8284363. Epub 2017 Oct 31. PMID 29226150
- [Background] Kupiec A, Zwierzchowski J, Kowal-Janicka J, Gozdzik W, Fuchs T, Pomorski M, Zimmer M, Kubler A. The analgesic efficiency of transversus abdominis plane (TAP) block after caesarean delivery. Ginekol Pol. 2018;89(8):421-424. doi: 10.5603/GP.a2018.0072. PMID 30215460
- [Background] Abdallah FW, Halpern SH, Margarido CB. Transversus abdominis plane block for postoperative analgesia after Caesarean delivery performed under spinal anaesthesia? A systematic review and meta-analysis. Br J Anaesth. 2012 Nov;109(5):679-87. doi: 10.1093/bja/aes279. Epub 2012 Aug 19. PMID 22907337
- [Background] Kwikiriza A, Kiwanuka JK, Firth PG, Hoeft MA, Modest VE, Ttendo SS. The analgesic effects of intrathecal morphine in comparison with ultrasound-guided transversus abdominis plane block after caesarean section: a randomised controlled trial at a Ugandan regional referral hospital. Anaesthesia. 2019 Feb;74(2):167-173. doi: 10.1111/anae.14467. Epub 2018 Nov 1. PMID 30383289
- [Background] Mishriky BM, George RB, Habib AS. Transversus abdominis plane block for analgesia after Cesarean delivery: a systematic review and meta-analysis. Can J Anaesth. 2012 Aug;59(8):766-78. doi: 10.1007/s12630-012-9729-1. Epub 2012 May 24. PMID 22622954